CLINICAL TRIAL: NCT00186797
Title: Purified CD34+ Hematopoietic Stem Cell Transplantation From Alternate Donors for Patients With Severe Aplastic Anemia
Acronym: AACD34
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AACD34
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Aplastic Anemia
Keywords: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — fludarabine; Cyclophosphamide

INTERVENTIONS:
Procedure: Allogeneic stem cell transplant
Drug: Fludarabine, Cyclophosphamide

SUMMARY:
This study is for patients with Severe Aplastic Anemia (SAA). A stem cell transplant from a genetically matched sibling donor can help or cure this disease in 85 to 100 percent of patients. Stem cells are immature blood cells that grow to become red blood cells, white blood cells or platelets. A genetic "match" means a brother or sister has same immune type (HLA type) as the patient. Unfortunately, few patients have a matched sibling donor. The chance of negative outcomes is much higher with other types of donors.

This study will test the success of a new approach to stem cell transplant for SAA. Patients in this study will receive drugs and radiation treatment to destroy their diseased bone marrow and to prepare them for stem cell transplant. Bone marrow is the tissue inside the bones where stem cells are made.Stem cells will be harvested from the blood or bone marrow of genetically matched unrelated donors or partially matched family donors. The stem cells will be filtered using a new device that is currently under study. The patients will receive large doses of the filtered stem cells (stem cell graft). Researchers want to find out how the study treatment affects patients, the disease, and the chances for survival.

ELIGIBILITY:
Inclusion Criteria:

* Age < 21 years
* Diagnosis of severe aplastic anemia. (As defined by at least 2 of the following: ANC < 500/μl, platelet count < 20,000/μl, and a reticulocyte count < 1% after correction for the hematocrit. In addition, the diagnostic bone marrow biopsy must contain less than 25% of the normal cellularity).
* Patient must have failed one or more courses of immunosuppressive therapy that included ATG. As immunosuppression may take up to 6 months to demonstrate a response, patients must have been observed to have failed immunosuppression for a minimum of six months.
* Absence of suitable HLA-matched sibling donor.
* Negative serum pregnancy test for females with child bearing potential.
* Patient/parent/guardian is able to provide informed consent.

Exclusion Criteria:

* Patients with a life expectancy < 6 weeks.
* Patients with severe renal disease (creatinine clearance < 40cc/min/1.73m2)
* Patients with pre-existing severe restrictive pulmonary disease (FVC <40% of predicted)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28
Dates: Start 2002-12; Primary Completion 2005-09 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To learn the safety of stem cell transplantation in patients with unrelated donors or partially matched family donors
To study the effects (good and bad) of this treatment on the patients, the aplastic anemia, and survival
To learn how well the donor bone marrow grows in patients who receive the research treatment
To learn how many patients need extra T-cells or extra stem cells from the donor to help the donor's blood stem cells grow

CONTACTS AND LOCATIONS:
Overall Officials: Paul Woodard, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org